CLINICAL TRIAL: NCT05519163
Title: A Study on Predictive Model for New-onset Diabetic Foot in Type 2 Diabetes Patients: A Retrospective Cohort Study.
Brief Title: A Study on Predictive Model for New-onset Diabetic Foot in Type 2 Diabetes Patients.
Status: Completed | Type: Observational
Sponsor: Yibing Wang (Other)
Responsible Party: Sponsor-Investigator, Yibing Wang, professor, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: YXLL-KY-2022(063)
Record Dates: First submitted 2022-08-26; First posted 2022-08-29 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Diabetic Foot
Keywords: Diabetes Mellitus, Type 2; Diabetic Foot; Predictive model; cohort study
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with type 2 diabetes: Patients with type 2 diabetes who were hospitalized in The First Affiliated Hospital of Shandong First Medical University & Shandong Provincial Qianfoshan Hospital between January 1, 2016 and December 31, 2021.

SUMMARY:
A retrospective cohort study was constructed based on hospitalized patients with type 2 diabetes, aiming to explore the related factors for new-onset diabetic foot and conducted a robust prediction model by Cox proportional hazards model.

DETAILED DESCRIPTION:
Diabetic foot is an infection of lower extremity, ulceration and/or deep tissue damage due to neuropathy and varying degrees of vascular disease in diabetic patients, including diabetic foot ulcerations or infections. Diabetic foot can lead to adverse consequences such as amputation and death,which seriously endangering the physical and mental health and quality of life for patients. Early identification of risk factors for diabetes foot is useful to reduce the risk of hospitalization, amputation or even mortality.

Most prediction models for diabetic foot focus on recurrent diabetic foot, however there is little published information on new-onset diabetic foot. This study aims to conduct a retrospective cohort based on Shandong Provincial Qianfoshan Hospital Healthcare Big Data Platform and build a prediction model for the new-onset diabetic foot using the related risk factors, which is of guidance significance for clinical prevention and treatment of diabetic foot.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of type 2 diabetes
2. Hospitalized patients
3. The interval between two records is more than one year

Exclusion Criteria:

1. Any history of ulcer or amputation previously
2. The patients with type 1 diabetes
3. Pregnant during the study
4. Patients with malignant tumors
5. Complicated with serious organ dysfunction, such as heart, liver and kidney

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with type 2 diabetes who were hospitalized in The First Affiliated Hospital of Shandong First Medical University & Shandong Provincial Qianfoshan Hospital between January 1, 2016 and December 31, 2021.
Sampling Method: Non-Probability Sample
Enrollment: 6301 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
New-onset diabetic foot | through study completion, an average of 32 months
  Diabetic foot was defined based on the self-reported disease history and clinical diagnosis from the electronic medical records. New-onset diabetic foot was diagnosed as the first-episode during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Wang Yibing, Doctor, Principal Investigator — The First Affiliated Hospital of Shandong First Medical University & Shandong Provincial Qianfoshan Hospital
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University & Shandong Provincial Qianfoshan Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Li MZ, Tang F, Liu YF, Lao JH, Yang Y, Cao J, Song R, Wu P, Wang YB. Risk factors and a predictive model of diabetic foot in hospitalized patients with type 2 diabetes. World J Diabetes. 2025 Mar 15;16(3):95644. doi: 10.4239/wjd.v16.i3.95644. PMID 40093275